CLINICAL TRIAL: NCT03945175
Title: Study of the Duration and Efficacy of MYDAYIS on Adult ADHD Symptoms and Executive Function Throughout the Day Into the Early Evening
Acronym: MYDAYIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00046
Record Dates: First submitted 2019-05-06; First posted 2019-05-10 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Attention Deficit-Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): After a two-week, single-blinded, placebo lead-in, all patients will receive four weeks of order-fixed treatment with Mydayis.
  Interventions: Drug: MYDAYIS; Drug: Placebo

INTERVENTIONS:
Drug: MYDAYIS — MYDAYIS treatment will be given at a minimum dose of 12.5mg/day and will increase in increments of 12.5mg, up to 37.5mg, based upon clinical response and tolerability.
Drug: Placebo — During the two-week, placebo lead-in, all patients will receive 12.5mg of placebo at Visit 1 and Visit 2.

SUMMARY:
Attention-deficit/hyperactivity disorder (ADHD) is a neuropsychiatric disorder characterized by problems with sustaining attention, organization, planning, procrastination, daydreaming, restlessness, impulsivity and hyperactivity.This is an outpatient study for subjects between the ages of 18-60, who have an Attention deficit hyperactivity disorder (ADHD) diagnosis meeting all inclusion criteria and not meeting any of the exclusion criteria.

DETAILED DESCRIPTION:
One purpose of this trial is to extend the evidence basis for Mydayis in adult ADHD to include efficacy with a clinical ADHD symptom measure validated for DSM-5 adult ADHD. Another purpose of this trial is to re-examine the clinical efficacy of Mydayis later in the day on ADHD symptoms; the data on ADHD symptoms via the TASS 1 (Spencer et al. 2008) is a decade old and has not been examined in subsequent trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18-60 of all races and ethnicity.
* Meets DSM V-TR criteria for a primary diagnosis of ADHD (including predominantly inattentive presentation, or combined presentation) as diagnosed via the Adult ADHD Clinician Diagnostic Scale version 1.2 (ACDS v1.2)

Exclusion Criteria:

* Meets DSM V-TR criteria for a primary diagnosis of hyperactive-impulsive type ADHD as diagnosed via the ACDS v1.2.
* Any other current psychiatric disorder, determined via the M.I.N.I, which requires pharmacotherapy treatment.
* Current suicidal ideation or history of suicide attempts, based on the Columbia- Suicide Severity Rating Scale(C-SSRS)
* Lifetime history of bipolar disorder or any psychotic disorder as per the M.I.N.I
* Pregnant, breastfeeding or women planning to become pregnant.
* Positive urine drug toxicology are excluded.
* Any other reason that, in the opinion of the investigator, prevents the subject from participating in the study or compromise the subject safety.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lenard Adler, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Then Mydayis: After a two-week, single-blinded, placebo lead-in, all patients will receive four weeks of order-fixed treatment with Mydayis.
  MYDAYIS: MYDAYIS treatment will be given at a minimum dose of 12.5mg/day and will increase in increments of 12.5mg, up to 37.5mg, based upon clinical response and tolerability.
  Placebo: During the two-week, placebo lead-in, all patients will receive 12.5mg of placebo at Visit 1 and Visit 2.
Period: Overall Study
Arm/Group | Placebo, Then Mydayis
Started (Participants Assessed for Eligibility) | 52
Participants Who Met Inclusion Criteria | 21
Participants Allocated to Single-Blind Placebo Treatment | 21
Participants Who Completed Single-Blind Placebo Treatment | 20
Participants Allocated to Mydayis Treatment | 18
Participants Included in Analysis of Outcome Measures | 18
Completed | 17
Not Completed | 35
Not completed — Did not meet inclusion criteria | 31
Not completed — Withdrew consent | 2
Not completed — Responded to Placebo Treatment and was not Allocated to Mydayis | 1
Not completed — Early termination during Mydayis treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Adult ADHD Investigator Symptom Rating Scale (AISRS) Score at End of Placebo Lead-In
Description: 18-item questionnaire measuring aspects of ADHD in adults. Participants rank items on a 4-point Likert scale: 0 (none), 1 (mild), 2 (moderate), 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of ADHD.
Time Frame: Week 2 (End of Placebo Lead-In)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 37.2 (11.4)

2. Primary Outcome: Adult ADHD Investigator Symptom Rating Scale (AISRS) Score at End of Mydayis Treatment
Description: as for outcome 1
Time Frame: Week 6 (End of Mydayis Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 18.5 (8.9)

3. Secondary Outcome: AISRS: Overall Inattentive (IA) Symptom Subscale Score at End of Placebo Lead-In
Description: The IA symptom subscale comprises 9 items of the AISRS measuring inattentive symptoms of ADHD. Items are ranked on a 4-point Likert scale: 0 (none), 1 (mild), 2 (moderate), 3 (severe). The total IA subscale score ranges from 0 to 27; higher scores indicate more severe IA symptoms.
Time Frame: Week 2 (End of Placebo Lead-In)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 19.9 (6.1)

4. Secondary Outcome: AISRS: Overall Inattentive (IA) Symptom Subscale Score at End of Mydayis Treatment
Description: as for outcome 3
Time Frame: Week 6 (End of Mydayis Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 9.6 (4.7)

5. Secondary Outcome: AISRS: Hyperactive-Impulsive (HI) Symptom Subscale Score at End of Placebo Lead-In
Description: The HI symptom subscale comprises 9 items of the AISRS measuring hyperactive-impulsive symptoms of ADHD. Items are ranked on a 4-point Likert scale: 0 (none), 1 (mild), 2 (moderate), 3 (severe). The total IA subscale score ranges from 0 to 27; higher scores indicate more severe HI symptoms.
Time Frame: Week 2 (End of Placebo Lead-In)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 17.3 (5.8)

6. Secondary Outcome: AISRS: Hyperactive-Impulsive (HI) Symptom Subscale Score at End of Mydayis Treatment
Description: as for outcome 5
Time Frame: Week 6 (End of Mydayis Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 8.8 (5.0)

7. Secondary Outcome: Clinical Global Impression-Severity (CGI-S) Scale Score at End of Placebo Lead-In
Description: 7-item questionnaire requiring a clinician to rate the severity of a patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. The ratings range from 1-7, where: 1 = Normal, not at all ill; 2 = Borderline mentally ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; and 7 = Among the most extremely ill patients.
Time Frame: Week 2 (End of Placebo Lead-In)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 4.6 (0.8)

8. Secondary Outcome: Clinical Global Impression-Severity (CGI-S) Scale Score at End of Mydayis Treatment
Description: as for outcome 7
Time Frame: Week 6 (End of Mydayis Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 3.1 (1.0)

9. Secondary Outcome: 14-Hour Post-Dose Time-Sensitive Adult ADHD Symptom Scale (TASS) Score at End of Placebo Lead-In
Description: 18-item assessment of the severity of ADHD symptoms administered 14 hours after morning dosing. Items are ranked on a 4-point Likert scale: 0 (not at all), 1 (mild), 2 (moderate), 3 (severe). The total score is the sum of all the items on the scale and ranges from 0 to 54. A higher total score indicates more severe ADHD.
Time Frame: Week 2 (End of Placebo Lead-In)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 24.6 (10.8)

10. Secondary Outcome: 14-Hour Post-Dose Time-Sensitive Adult ADHD Symptom Scale (TASS) Score at End of Mydayis Treatment
Description: as for outcome 9
Time Frame: Week 6 (End of Mydayis Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 16.8 (10.8)

11. Secondary Outcome: 14-hour Post-Dose TASS: Inattentive (IA) Symptom Subscale Score at End of Placebo Lead-In
Description: The IA symptom subscale comprises 9 items of the TASS measuring inattentive symptoms of ADHD. Items are ranked on a 4-point Likert scale: 0 (not at all), 1 (mild), 2 (moderate), 3 (severe). The total IA subscale score ranges from 0 to 27; higher scores indicate more severe IA symptoms. Administered 14 hours after morning dosing.
Time Frame: Week 2 (End of Placebo Lead-In)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 15.4 (5.5)

12. Secondary Outcome: 14-hour Post-Dose TASS: Inattentive (IA) Symptom Subscale Score at End of Mydayis Treatment
Description: as for outcome 11
Time Frame: Week 6 (End of Mydayis Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 9.8 (6.3)

13. Secondary Outcome: 14-hour Post-Dose TASS: Hyperactive-Impulsive (HI) Symptom Subscale Score at End of Placebo Lead-In
Description: The HI symptom subscale comprises 9 items of the TASS measuring inattentive symptoms of ADHD. Items are ranked on a 4-point Likert scale: 0 (not at all), 1 (mild), 2 (moderate), 3 (severe). The total IA subscale score ranges from 0 to 27; higher scores indicate more severe HI symptoms. Administered 14 hours after morning dosing.
Time Frame: Week 2 (End of Placebo Lead-In)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 9.2 (5.7)

14. Secondary Outcome: 14-hour Post-Dose TASS: Hyperactive-Impulsive (HI) Symptom Subscale Score at End of Mydayis Treatment
Description: as for outcome 13
Time Frame: Week 6 (End of Mydayis Treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 6.9 (5.3)

15. Secondary Outcome: Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Score at Week 3
Description: 75-item questionnaire measuring an adult's cognitive, emotional, and behavioral functions within the past month. Items ranked on 3-point Likert scale (1 = Never, 2 = Sometimes, 3 = Often). Raw scores are calculated and used to generate T-scores for 8 scales (Inhibit; Shift; Emotional Control; Initiate; Working Memory; Plan/Organize; Task Monitor; and Organization of Materials), 2 summary index scales (Behavioral Regulation Index and Metacognition Index), and 1 scale reflecting overall functioning (Global Executive Composite). T-scores range from 30 to 100, with scores ≥65 indicating clinical impairment.
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
T-score | 68.6 (8.9)

16. Secondary Outcome: Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) Score at Week 7
Description: as for outcome 15
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
T-score | 58.6 (14.9)

17. Secondary Outcome: WebNeuro Neurocognitive Assessment - Working Memory Capacity - Recall Span Score at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the working memory capacity - recall span domain, participants complete forward digit span task and are assessed based on the maximum length of a sequence of visually presented digits able to be entered on a keypad in correct order. The total score is the maximum length of the sequence of digits.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: digits
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
digits | 5.8 (2.0)

18. Secondary Outcome: WebNeuro Neurocognitive Assessment - Working Memory Capacity - Recall Span Score at Week 7
Description: as for outcome 17
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
score on a scale | 6.4 (1.2)

19. Secondary Outcome: WebNeuro Neurocognitive Assessment - Working Memory Capacity - Working Memory Accuracy at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the working memory capacity - working memory accuracy domain, participants complete a digit span task. Participants are assessed based on the total number of correct trials in the forward digit span task where each incremental span length has two trials- at least one of which needs to be recalled correctly to progress.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: trials correct
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
trials correct | 6.9 (3.2)

20. Secondary Outcome: WebNeuro Neurocognitive Assessment - Working Memory Capacity - Working Memory Accuracy at Week 7
Description: as for outcome 19
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: trials correct
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
trials correct | 7.7 (2.1)

21. Secondary Outcome: WebNeuro Neurocognitive Assessment - Attention and Concentration - Reaction Time at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the attention and concentration - reaction time domain, participants complete a continuous performance test. Participants are assessed based on their reaction time to space-bar presses, averaged across all correctly identified target stimuli (same letter presented twice in a row).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 567.0 (118.0)

22. Secondary Outcome: WebNeuro Neurocognitive Assessment - Attention and Concentration - Reaction Time at Week 7
Description: as for outcome 21
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 566.3 (145.4)

23. Secondary Outcome: WebNeuro Neurocognitive Assessment - Attention and Concentration - False Alarms at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the attention and concentration - false alarms domain, participants complete a continuous performance test. Participants are assessed based on the number of times the space-bar was pressed at any time not in response to a "target" stimulus.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of false alarms
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of false alarms | 1.3 (1.2)

24. Secondary Outcome: WebNeuro Neurocognitive Assessment - Attention and Concentration - False Alarms at Week 7
Description: as for outcome 23
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of false alarms
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of false alarms | 1.0 (1.3)

25. Secondary Outcome: WebNeuro Neurocognitive Assessment - Attention and Concentration - False Misses at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the attention and concentration - false misses domain, participants complete a continuous performance test. Participants are assessed based on the number of times when the space-bar was NOT pressed following a target stimulus.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of false misses
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of false misses | 0.7 (0.9)

26. Secondary Outcome: WebNeuro Neurocognitive Assessment - Attention and Concentration - False Misses at Week 7
Description: as for outcome 25
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of false misses
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of false misses | 0.7 (1.0)

27. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Completion Time at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the information processing efficiency - completion time domain, participants complete a switching of attention task. Participants are assessed based on the total amount of time taken to complete the whole sequence of digits and letters.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 56771.9 (12548.0)

28. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Completion Time at Week 7
Description: as for outcome 27
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 47752.6 (12867.6)

29. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Average Connection Time at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the information processing efficiency - average connection time domain, participants complete a switching of attention task. Participants are assessed based on the average time between correct responses.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 2228.0 (617.3)

30. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Average Connection Time at Week 7
Description: as for outcome 29
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 1863.1 (517.9)

31. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Errors at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the information processing efficiency - errors domain, participants complete a switching of attention task. Participants are assessed based on the number of times an incorrect digit or letter in the sequence was pressed.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of errors
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of errors | 0.8 (1.2)

32. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Errors at Week 7
Description: as for outcome 31
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of errors
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of errors | 0.7 (0.7)

33. Secondary Outcome: WebNeuro Neurocognitive Assessment - Response Speed - Number of Taps at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the response speed - number of taps domain, participants complete a motor tapping task. Participants are assessed based on the number of times they were able to tap the spacebar in 30 seconds with their dominant hand.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of taps
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of taps | 189.6 (22.2)

34. Secondary Outcome: WebNeuro Neurocognitive Assessment - Response Speed - Number of Taps at Week 7
Description: as for outcome 33
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of taps
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of taps | 189.9 (20.0)

35. Secondary Outcome: WebNeuro Neurocognitive Assessment - Response Speed - Tapping Variability at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the response speed - tapping variability domain, participants complete a motor tapping task. Participants are assessed based on the standard deviation of the time interval between taps on the space-bar for the dominant hand.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 24.4 (7.8)

36. Secondary Outcome: WebNeuro Neurocognitive Assessment - Response Speed - Tapping Variability at Week 7
Description: as for outcome 35
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 30.4 (24.2)

37. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Reaction Time at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the information processing efficiency - reaction time domain, participants complete a choice reaction time task. Participants are assessed based on the average time taken to press the left or right arrow to correspond with which circle (left or right) is highlighted in each trial.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 379.2 (38.5)

38. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Reaction Time at Week 7
Description: as for outcome 37
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 378.2 (48.7)

39. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Score (Words) at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the information processing efficiency - score (words) domain, participants complete a verbal interference (word) task. Participants are assessed based on the number of stimuli for which the name of the color-word was correctly selected (ignoring the font-color of the word) in the time limit of 30 seconds (i.e., a higher score reflects greater speed).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of correct trials
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of correct trials | 15.4 (5.1)

40. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Score (Words) at Week 7
Description: as for outcome 39
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of correct trials
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of correct trials | 16.0 (4.0)

41. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Errors (Words) at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the information processing efficiency - errors (words) domain, participants complete a verbal interference (word) task. Participants are assessed based on the number of stimuli for which the name of the color-word was incorrectly selected (ignoring the font-color of the word) in the time limit of 30 seconds (i.e., a higher score reflects more errors).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of incorrect trials
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of incorrect trials | 0.2 (0.8)

42. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Errors (Words) at Week 7
Description: as for outcome 41
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of incorrect trials
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of incorrect trials | 0.4 (1.2)

43. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Reaction Time (Words) at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the information processing efficiency - reaction time (words) domain, participants complete a verbal interference (word) task. Participants are assessed based on the average reaction time for the stimuli for which the name of the color-word was correctly selected (ignoring the font-color of the word).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 1434.5 (961.6)

44. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Reaction Time (Words) at Week 7
Description: as for outcome 43
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 1248.4 (315.2)

45. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Score (Colors) at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the information processing efficiency - score (colors) domain, participants complete a verbal interference (color) task. Participants are assessed based on the number of stimuli for which the font-color of the color-word was correctly selected (ignoring the name of the word) in the time limit of 30 seconds (i.e., a higher score reflects greater speed).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of correct trials
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of correct trials | 12.8 (4.2)

46. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Score (Colors) at Week 7
Description: as for outcome 45
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of correct trials
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of correct trials | 15.7 (4.9)

47. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Errors (Colors) at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the information processing efficiency - errors (colors) domain, participants complete a verbal interference (color) task. Participants are assessed based on the number of stimuli for which the font-color of the color-word was incorrectly selected (ignoring the name of the word) in the time limit of 30 seconds (i.e., a higher score reflects more errors).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of incorrect trials
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of incorrect trials | 0.3 (0.8)

48. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Errors (Colors) at Week 7
Description: as for outcome 47
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of incorrect trials
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of incorrect trials | 2.1 (7.0)

49. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Reaction Time (Colors) at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the information processing efficiency - reaction time (colors) domain, participants complete a verbal interference (color) task. Participants are assessed based on the average reaction time for the stimuli for which the font-color of the color-word was correctly selected (ignoring the name of the word).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 1526.8 (399.2)

50. Secondary Outcome: WebNeuro Neurocognitive Assessment - Information Processing Efficiency - Reaction Time (Colors) at Week 7
Description: as for outcome 49
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 1176.2 (263.7)

51. Secondary Outcome: WebNeuro Neurocognitive Assessment - Executive Function - Trials Completed at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the executive function - trials completed domain, participants complete a maze task. Participants are assessed based on the number of trials taken to successfully complete the maze without error twice consecutively.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of trials completed
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of trials completed | 9.5 (4.8)

52. Secondary Outcome: WebNeuro Neurocognitive Assessment - Executive Function - Trials Completed at Week 7
Description: as for outcome 51
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of trials completed
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of trials completed | 8.1 (3.9)

53. Secondary Outcome: WebNeuro Neurocognitive Assessment - Executive Function - Completion Time at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the executive function - completion time domain, participants complete a maze task. Participants are assessed based on the time taken to successfully complete the maze without error twice consecutively.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 234774.9 (87879.2)

54. Secondary Outcome: WebNeuro Neurocognitive Assessment - Executive Function - Completion Time at Week 7
Description: as for outcome 53
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 174054.1 (93675.1)

55. Secondary Outcome: WebNeuro Neurocognitive Assessment - Executive Function - Path Learning Time at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the executive function - path learning time domain, participants complete a maze task. Participants are assessed based on the time taken to the end of the final trial with at least one error- just before successfully completing the maze without error twice consecutively.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 204859.7 (81156.1)

56. Secondary Outcome: WebNeuro Neurocognitive Assessment - Executive Function - Path Learning Time at Week 7
Description: as for outcome 55
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 148589.5 (88469.0)

57. Secondary Outcome: WebNeuro Neurocognitive Assessment - Executive Function - Total Errors at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the executive function - total errors domain, participants complete a maze task. Participants are assessed based on the cumulative number of all types of errors made across all trials taken to complete the maze without error twice consecutively.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of incorrect moves
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of incorrect moves | 37.1 (27.0)

58. Secondary Outcome: WebNeuro Neurocognitive Assessment - Executive Function - Total Errors at Week 7
Description: as for outcome 57
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of incorrect moves
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of incorrect moves | 26.3 (13.1)

59. Secondary Outcome: WebNeuro Neurocognitive Assessment - Executive Function - Number of Overruns at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the executive function - number of overruns domain, participants complete a maze task. Participants are assessed based on the cumulative number of 'overrun' errors made across all trials taken to complete the maze without error twice consecutively. Overrun errors are specifically when subjects continue pressing in the same direction of movement through the maze instead of turning where required.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of incorrect moves
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of incorrect moves | 14.8 (14.8)

60. Secondary Outcome: WebNeuro Neurocognitive Assessment - Executive Function - Number of Overruns at Week 7
Description: as for outcome 59
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of incorrect moves
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of incorrect moves | 12.8 (7.3)

61. Secondary Outcome: WebNeuro Neurocognitive Assessment - Impulsivity - Reaction Time at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the impulsivity - reaction time domain, participants complete a Go/No-Go task. Participants are assessed based on reaction time to spacebar press averaged across all correctly performed green "press" stimuli.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 308.2 (63.6)

62. Secondary Outcome: WebNeuro Neurocognitive Assessment - Impulsivity - Reaction Time at Week 7
Description: as for outcome 61
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
milliseconds | 307.8 (48.2)

63. Secondary Outcome: WebNeuro Neurocognitive Assessment - Impulsivity - False Alarms at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the impulsivity - false alarms domain, participants complete a Go/No-Go task. Participants are assessed based on the number of times when the spacebar was pressed at any time in response to a red "don't press" stimulus.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Number of spacebar presses
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of spacebar presses | 6.1 (3.5)

64. Secondary Outcome: WebNeuro Neurocognitive Assessment - Impulsivity - False Alarms at Week 7
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the impulsivity - false alarms domain, participants complete a Go/No-Go task. Participants are assessed based on the number of times when the spacebar was pressed a1t any time in response to a red "don't press" stimulus.
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of spacebar presses
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of spacebar presses | 5.2 (3.6)

65. Secondary Outcome: WebNeuro Neurocognitive Assessment - Impulsivity - False Misses at Baseline
Description: WebNeuro is a web-based computerized battery of several domains of neurocognitive functioning. In the impulsivity - false misses domain, participants complete a Go/No-Go task. Participants are assessed based on the number of times when the spacebar was not pressed in response to a green "press" stimulus.
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of spacebar presses
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of spacebar presses | 1.9 (2.0)

66. Secondary Outcome: WebNeuro Neurocognitive Assessment - Impulsivity - False Misses at Week 7
Description: as for outcome 65
Time Frame: Week 7
Measure: Mean (Standard Deviation); unit: Number of spacebar presses
Arm/Group | Placebo, Then Mydayis
Number analyzed (Participants) | 18
Number of spacebar presses | 0.3 (0.6)

ADVERSE EVENTS:
Time Frame: 7 Weeks
Description: Participants monitored weekly for abnormal vital signs, adverse events, and concomitant medications.
Arm/Group | Placebo, Then Mydayis
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 14/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo, Then Mydayis (N=18)
Headache (Nervous system disorders) | 5
Pain - Arm (General disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Allergic Reaction (Immune system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Burn (Injury, poisoning and procedural complications) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Tachycardia (Cardiac disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 1
COVID-19 (General disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 2
Other - Increased Appetite (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Pain - Foot (General disorders) | 1
Agitation (Psychiatric disorders) | 1
Concentration impairment (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-02): https://cdn.clinicaltrials.gov/large-docs/75/NCT03945175/Prot_SAP_000.pdf